CLINICAL TRIAL: NCT06526195
Title: Trial to Evaluate Safety And Effectiveness of Mechanical Circulatory Support in Patients With Advancing Heart Failure
Acronym: TEAM-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT- CIP-10521
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Heart Diseases; Cardiovascular Diseases; Pulmonary Hypertension
Keywords: Heart Failure; Left Ventricular Assist Device (LVAD); Guideline Directed Medical Therapy (GDMT); Non-inotrope Dependent; Pulmonary Artery Pressure; Hemodynamic Monitoring; Medical Management; CardioMEMS; HeartMate 3 (HM3); Ambulatory Advanced Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Randomized Arm - HM3 Group (Experimental): Patients with elevated mean PAP (mean PAP ≥ 30 mmHg) and randomized to the HM3 group will receive the device within 14 days of randomization.
  Interventions: Device: CardioMEMS HF System; Device: HeartMate 3 Left Ventricular Assist System; Other: Guideline Medical Directed Therapy
- Randomized Arm - Control Group (Experimental): Patients with elevated mean PAP (mean PAP ≥ 30 mmHg) and randomized to the control group will continue their medical therapy per established heart failure guidelines.
  Interventions: Device: CardioMEMS HF System; Other: Guideline Medical Directed Therapy
- Single Arm Registry (Experimental): Patients who do not meet the mean PAP threshold (mean PAP <30 mmHg) and are enrolled in the single arm will continue their medical therapy per established heart failure guidelines.
  Interventions: Device: CardioMEMS HF System; Other: Guideline Medical Directed Therapy

INTERVENTIONS:
Device: CardioMEMS HF System — The CardioMEMS™ HF System is comprised of a lead-less and battery-less pressure sensor which remotely transmits pulmonary artery pressure measurements.
  Other Names: CardioMEMS; CardioMEMS PA Sensor
Device: HeartMate 3 Left Ventricular Assist System — The HeartMate 3 LVAS is a mechanical circulatory support pump with Full MagLev Technology that assumes some or all of the workload of the left ventricle. The HeartMate 3 LVAS is used in advanced heart failure patients needing short or long-term mechanical circulatory support.
  Other Names: HM3
  Arms: Randomized Arm - HM3 Group
Other: Guideline Medical Directed Therapy — Optimal doses of medical therapy per established heart failure guidelines which includes the following stable combination of Beta Blockers, ACE-inhibitors or ARB or ARNi, MRA and SGLT2 inhibitors.
  Other Names: GDMT

SUMMARY:
The purpose of TEAM-HF IDE clinical trial is to evaluate safety and effectiveness of the HeartMate 3 LVAS compared to guideline directed medical therapy (GDMT) in a population of ambulatory advanced heart failure patients who are not dependent on intravenous inotrope.

DETAILED DESCRIPTION:
Patients with heart failure (HF) suffer from a high degree of morbidity and mortality. Left ventricular assist device (LVAD) therapy has become the standard of care for the treatment of advanced HF patients who are deemed to be dependent on continuous intravenous inotropes, extending life expectancy, enhancing overall quality of life, and improving functional capacity. However, use of LVADs in ambulatory, non-inotrope dependent advanced HF population is limited. Elevated mean pulmonary artery pressure (PAP) secondary to left ventricular failure has emerged as a potential predictor of increased mortality risk for patients refractory to maximally tolerated guideline directed medical therapy (GDMT). In these patients, left ventricular failure with elevated mean PAP may represent objective criteria to identify advanced HF patients requiring heart replacement therapies such as LVAD.

The TEAM-HF IDE trial will enroll approximately 850 subjects with New York Heart Association (NYHA) Class IIIB/IV HF who had a prior heart failure hospitalization and an elevated mean PAP secondary to left ventricular failure. Elevated mean PAP will be identified using an implanted PAP monitoring sensor, the CardioMEMS PA Sensor. All subjects enrolled can have a previously implanted CardioMEMS PA Sensor or, if not, will be implanted with the CardioMEMS PA Sensor after enrollment. The overall objectives of TEAM-HF trial are two-fold: 1) To determine whether PAP can objectively identify patients most at risk for worsening HF and therefore most likely to benefit from earlier intervention with LVAD therapy and 2) To determine the benefit of LVAD therapy in non-inotrope advanced HF patients with elevated mean PAP refractory to GDMT.

The trial will include approximately 75 global sites and consists of a Randomized Arm and a Single Arm Registry.

The TEAM-HF Randomized Arm is a prospective, randomized, open-label study of the HeartMate 3 (HM3) left ventricular assist system (LVAS) versus continued GDMT in non-inotrope dependent HF patients. The objectives of the Randomized Arm are 1) To establish an objective disease-state criteria to trigger referral for a HM3 LVAS and 2) Demonstrate improvement in survival when non-inotrope dependent advanced HF patients are treated with the HM3 LVAS compared to being managed on medical therapy alone.

The TEAM-HF Single Arm Registry is a prospective, single-arm, open-label study of non-inotrope dependent HF patients who do not meet a mean PAP threshold after GDMT optimization. The objective of the Single Arm Registry is to characterize the progression of patients with non-inotrope dependent HF without elevated PAP.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent by signing the study Informed Consent Form (ICF) prior to any clinical investigation-related procedure
2. LVEF ≤30% and Cardiac Index ≤ 2.5 L/min/m²
3. Limited functional status as demonstrated by 6MWT ≤ 350 m due to HF related reasons OR peak VO2 ≤ 14 mL/kg/min (or <50% of predicted peak VO2 value)
4. NYHA Class IIIB or NYHA Class IV
5. Subject has ≥ 1 Heart Failure Hospitalization in the last 12 months
6. Subject is already implanted with a CardioMEMS PA Sensor OR willing to undergo a CardioMEMS PA Sensor implant
7. Subject is willing and able to be implanted with the HM3 LVAS if randomized to HM3 Group

Randomization Criteria:

1. Subject has been implanted with a CardioMEMS PA Sensor for at least 90 days.
2. Subject is receiving guideline directed medical therapy with optimal doses (or documented medication contraindication or intolerance) of betablockers, Angiotensin-Converting-Enzyme-inhibitors or Angiotensin II Receptor Blockers or angiotensin receptor neprilysin inhibitor (if eligible), Mineralocorticoid Receptor Antagonists, Sodium-Glucose co-Transporter-2 (SGLT2) inhibitors, and diuretics for at least 30 of the last 90 days.
3. mean PAP ≥ 30 mmHg.
4. The subject will not be randomized if they have any other factor that represents inordinate risk for either continued GDMT or LVAD implant.

Single Arm Registry Criteria:

1. Subject has received a CardioMEMS PA Sensor implant following enrollment in the trial.
2. Subject is receiving guideline directed medical therapy with optimal doses (or documented medication contraindication or intolerance) of betablockers, Angiotensin-Converting-Enzyme-inhibitors or Angiotensin II Receptor Blockers or angiotensin receptor neprilysin inhibitor (if eligible), Mineralocorticoid Receptor Antagonists, Sodium-Glucose co-Transporter-2 (SGLT2) inhibitors, and diuretics for at least 30 of the last 90 days.
3. mean PAP <30 mmHg

Exclusion Criteria:

1. Subject is < 18 years of age at the time of informed consent.
2. Dependent on IV inotrope in the last 30 days.
3. Contra-indications to HM3 LVAS or CardioMEMS HF system.
4. Etiology of HF due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, or restrictive cardiomyopathy.
5. Technical obstacles to LVAD or CardioMEMS implantation which pose an inordinately high surgical risk, in the judgment of the implanter.
6. Existence of ongoing MCS.
7. Presence of mechanical aortic valve that will not be either converted to a bioprosthesis or oversewn at the time of LVAD implant.
8. History of any solid organ transplant.
9. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAS management.
10. Presence of an active, uncontrolled infection.
11. Complex congenital heart disease.
12. Currently Pregnant or capable of becoming Pregnant and Unwilling to Use Contraception with LVAD.
13. History of pulmonary embolism within 30 days prior to enrollment or history of recurrent (>1 episode) pulmonary embolism and/or deep vein thrombosis.
14. Planned VAD or Bi-VAD support prior to enrollment.
15. Presence of any one of the following risk factors for or indications of severe end organ dysfunction or failure:

    1. An INR ≥ 2.0 not due to anticoagulation therapy
    2. An eGFR < 30 mL/min/1.73 m2 and nonresponsive to diuretic therapy or receiving chronic dialysis.
    3. Biopsy proven liver cirrhosis.
    4. Need for chronic renal replacement therapy.
    5. History of severe chronic obstructive pulmonary disease (COPD) defined by Forced Expiratory Volume FEV1 < 30% predicted.
    6. History of cerebrovascular disease with significant (> 80%) uncorrected internal carotid stenosis.
    7. Significant peripheral vascular disease (PVD) accompanied by ischemic rest pain or extremity ulceration.
16. Any condition other than HF that could limit survival to less than 24 months.
17. Participation in any other clinical investigation with an active treatment arm that is likely to confound study results or affect the study outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Survival at 2 years free of disabling stroke, reoperation to replace the device, or worsening HF requiring listing for urgent heart transplantation or mechanical circulatory support, enrollment into hospice, or dependence on IV inotropes | 2 years
  The powered primary endpoint will be analyzed at 2 years following the Com-Nougue method and will be compared between the HM3 Group (HM3 LVAD) and the Control Group (GDMT) within the Intention-to-treat (ITT) population.

SECONDARY OUTCOMES:
Rate of Safety Outcomes at 1-year | 1 year
  The powered secondary endpoint of Rate of Safety Outcomes at 1-year will be evaluated within the Intention-to-treat (ITT) population against a pre-specified performance goal.
  Components consist of the following:
  1. Heart failure hospitalization
  2. Major Adverse Event (MAE) including:
     * Stroke
     * Non-surgical bleeding (>14 days post implant) requiring hospitalization
     * Renal failure requiring hospitalization
     * Driveline infection requiring hospitalization
Survival at 2 years | 2 years
  The powered secondary endpoint of survival at 2-years will be compared between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population.
Quality of life score assessed with the Kansas City Cardiomyopathy Questionnaire | 2 years
  The secondary endpoint of Quality-of-life score at 2-years will be compared between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population. Additionally, the secondary endpoint of Quality of life at 2-years will be descriptively compared between the Single Arm Registry and both the HM3 Group and Control Group of the Randomized Arm separately.
  The KCCQ scores are represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life. Improvement of KCCQ by at least 10 points is considered clinically significant.
Six-minute walk distance | 2 years
  The secondary endpoint of six-minute walk distance at 2-years will be compared between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population. Additionally, the secondary endpoint of six-minute walk distance at 2-years will be descriptively compared between the Single Arm Registry and both the HM3 Group and Control Group of the Randomized Arm separately.
Hospitalizations for HF and/or Urgent HF Visit | 2 years
  The secondary endpoint of Hospitalizations for HF and/or Urgent HF Visit at 2-years will be compared between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population. Additionally, the secondary endpoint of Hospitalizations for HF and/or Urgent HF Visit at 2-years will be descriptively compared between the Single Arm Registry and both the HM3 Group and Control Group of the Randomized Arm separately.
Days alive and outside of the hospital | 2 years
  The secondary endpoint of days alive and outside of the hospital at 2-years will be compared between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population. Additionally, the secondary endpoint of days alive and outside of the hospital at 2-years will be descriptively compared between the Single Arm Registry and both the HM3 Group and Control Group of the Randomized Arm separately.
All-cause hospitalizations | 2 years
  The secondary endpoint of all-cause hospitalizations at 2-years will be compared between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population. Additionally, the secondary endpoint of all-cause hospitalizations at 2-years will be descriptively compared between the Single Arm Registry and both the HM3 Group and Control Group of the Randomized Arm separately.
All adverse events (including all strokes) regardless of severity | 2 years
  The secondary endpoint of all adverse events (including all strokes) regardless of severity at 2-years will be compared between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population. Additionally, the secondary endpoint of all adverse events (including all strokes) regardless of severity at 2-years will be descriptively compared between the Single Arm Registry and both the HM3 Group and Control Group of the Randomized Arm separately.

OTHER OUTCOMES:
Finkelstein-Schoenfeld Win Ratio | 5 years
  The Finkelstein-Schoenfeld Win Ratio will be explored at 5 years as an additional analysis with the following hierarchy:
  1. Survival
  2. Days alive outside of the hospital
  3. Quality of Life assessed with the KCCQ (considered a tie if within 10 points)
  4. Functional Capacity (Six-minute walk distance)
  The Finkelstein-Schoenfeld Win Ratio will be analyzed between the HM3 Group and the Control Group within the Intention-to-treat (ITT) population. Additionally, the Finkelstein-Schoenfeld Win Ratio will be descriptively analyzed between the Single Arm and both the HM3 Group and Control Group of the Randomized Arm separately.
Survival free of urgent LVAD or transplant | 5 years
  This additional descriptive analysis at 5-years will be performed to evaluate the proportion of patients who are alive and free of device replacement or transplant in the HM3 Group compared to the Single Arm Registry (de novo implant or transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly O'Connell, PhD, Study Director — Abbott
Locations (59):
- United States (48):
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Sutter Medical Center, Sacramento, California
  - University of California at San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Shands at the University of Florida, Gainesville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Piedmont Augusta Hospital, Augusta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Advocate Health & Hospitals Corporation, Oakbrook Terrace, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - North Shore University Hospital, Manhasset, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Midlands, Columbia, South Carolina
  - The Stern Cardiovascular Foundation, Memphis, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - Baylor University Hospital, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist, Houston, Texas
  - UTHealth Memorial Hermann, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Aurora Medical Group, Milwaukee, Wisconsin
- AKH -Wien, Vienna, Vienna, Austria
- IKEM Prague, Prague, CBohmia, Czechia
- Rigshospitalet, Copenhagen, Copenhagen, Denmark
- Germany (3):
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Medizinische Hochschule Hannover, Hanover, Saxon
  - Deutsches Herzzentrum der Charité, Berlin, State of Berlin
- A.O.U. Citta della Salute e della Scienza di Torino, Turin, Piedmont, Italy
- Netherlands (2):
  - Erasmus MC - Thoraxcenter, Rotterdam, Holland
  - UMC Utrecht, Utrecht, Utrecht
- Saudi Arabia (2):
  - King Fahad Medical City, Riyadh, Riyadh Region
  - King Faisal Specialist Hospital, Riyadh, Riyadh Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TEAM-HF Clinical Trial Patient Information — https://www.cardiovascular.abbott/us/en/campaigns/team-hf.html